CLINICAL TRIAL: NCT01150149
Title: Evaluating Modes of Influenza Transmission Using a Human Challenge/Exposure Model
Brief Title: Evaluating Modes of Influenza Transmission Between Humans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding application unsuccessful
Sponsor: University of Nottingham (Other)
Collaborators: Imperial College London (Other); University College, London (Other); Retroscreen Virology Ltd. (Industry)
Responsible Party: Paul Cartledge, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08145
Record Dates: First submitted 2009-08-10; First posted 2010-06-24 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Influenza
Keywords: Influenza; Humans; Experimental; Challenge
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention)
- 2 (Experimental): No face touch
  Interventions: Behavioral: No face touch
- 3 (Experimental): Surgical face mask
  Interventions: Device: Surgical face mask
- 4 (Experimental): Surgical face mask + no face touch
  Interventions: Device: Surgical face mask + no face touch

INTERVENTIONS:
Behavioral: No face touch
  Arms: 2
Device: Surgical face mask
  Arms: 3
Device: Surgical face mask + no face touch
  Arms: 4

SUMMARY:
Most countries of the world, including the USA are making preparations for a possible influenza pandemic. Such an event will constitute a global public health emergency, but it is impossible to predict when this will happen. Up to 80 million people could die worldwide, so as much as possible needs to be done in advance to find ways of how the impact can be reduced. Although the investigators know that medical interventions such as anti-influenza drugs and antibiotics will be important, even in well resourced countries these might be in short supply. Vaccines will also be important but these will not be available until at least 4-5 months after the pandemic has started. This means that other non-pharmaceutical measures could well be important such as social distancing, school closures and the use of face masks. Guidance also needs to be developed so that families can care for each other whilst minimizing the spread of infection. To do these things, the investigators need to know how influenza is transmitted from person-to person. This is poorly understood at present. The investigators also need to know if face masks work before recommendations for public use can be made. The best way to study influenza transmission and the effectiveness of masks is to perform a study using healthy adult volunteers. The investigators will do this by giving some volunteers normal influenza via nasal drops. When they get symptoms the investigators will create an 'experimental household' by getting them to live with other non-infected volunteers for 48 hours, in a specially designed quarantine isolation unit. Some of the non-infected volunteers will be unprotected; others will be selected randomly to wear either face masks or a special plastic 'cloak' so that they do not touch their faces; another group will wear both. The investigators will then measure the rate at which the different groups get 'flu'. From these data the investigators can work out whether it is touching the face or coughing and sneezing that spreads flu most or whether both are important; the investigators can also deduce how well face masks work to prevent spread. The investigators need almost 2000 volunteers for this study, it will take at least 2 years to complete and it will be very costly, however, the results will be of global importance. If the study is successful, the investigators can tell governments around the world whether face masks work to prevent influenza and be clearer about the guidance that should be given to families.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive.
* Comprehension of the study requirements; availability for the required study period, ability to attend scheduled study visits, and willingness to participate in the inpatient challenge.
* Willingness to provide written consent for participation after reading the Subject Information Sheet and Informed Consent Form and after having adequate opportunity to discuss the study with an Investigator or qualified deputy.
* H3N2 antibody titre levels recorded as < 1:10
* Good general health status as determined by a screening evaluation no greater than 160 days prior to the quarantine challenge phase.
* Subjects shall be registered with a general practitioner who will confirm a subjects' past medical history and their suitability to participate based on this. Consent will be obtained to receive this information.
* For female subjects, provision of a history of reliable contraceptive practices [hysterectomy or bilateral tubal ligation, oral or implanted contraceptive use, intrauterine device, barrier method plus spermicide, history of a single male partner with vasectomy and documentary evidence confirming sterility (negative sperm counts at the recommended post-operative intervals) or a history of abstinence deemed credible by the Investigator]. The provision of this history does NOT replace the requirement to perform, and obtain negative results in, pregnancy tests.

Exclusion Criteria:

* Presence of any significant acute or chronic, uncontrolled medical or psychiatric illness, including but not exclusive to the conditions listed in Appendix 7, that in the view of the Investigator is associated with increased risk of complications of respiratory viral illness [subjects with uncomplicated chronic diagnoses stable and treated for 3 months (e.g. mild hypertension well-controlled with medication may be enrolled) provided the condition and its therapy are not known to be associated with an immunocompromised state or increased risk of complications of respiratory viral illness].
* Health care workers (including doctors, nurses, medical students and allied healthcare professionals) anticipated to have patient contact within two weeks of viral challenge. Healthcare workers who volunteer should not work with patients until 14 days after challenge or until their symptoms are fully resolved (whichever is the longer). Health care workers who work in units housing severely immunocompromised patients (e.g. bone marrow transplant units) will be excluded from the study.
* Venous access deemed inadequate for the phlebotomy demands of the study.
* Positive serologic tests for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
* Evidence of drug abuse or a positive urine Class A drug or alcohol screen.
* Female subjects, who are known to be pregnant or who have a positive urine pregnancy test prior to challenge.
* Acute (within 7 days of challenge/exposure) or chronic use of any medication or other product (prescription or over-the-counter), for symptoms of rhinitis or nasal congestion or for any nasopharyngeal complaint, or use of any intranasal medication for any indication (this includes any corticosteroid or beta agonist containing nasal spray).
* Any history during adulthood of asthma, chronic obstructive pulmonary disease or any other condition requiring bronchodilator therapy. A history of childhood asthma until and including the age of 12 is acceptable.
* Smokers unwilling/unable to desist for the quarantine phase duration of the study and any smoker who has a >10 pack year history of smoking. A nicotine test will be done at study specific screening and must be negative prior to admission to the quarantine unit.
* Subjects who have type I or type II Diabetes Mellitus.
* Body Mass Index > 30.
* An Abnormal ECG deemed clinically relevant by the Investigator.
* Any anatomic or neurologic abnormality impairing the gag reflex or conducive to aspiration, or history suggestive of such a problem or any abnormality significantly altering the anatomy of the nose or nasopharynx.
* Receipt of systemic glucocorticoids (in a dose 5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within six months prior to challenge.
* Receipt of any investigational drug within 6 months prior to challenge, or prior participation in a clinical trial of any Influenza vaccine, or any investigational vaccine or experimental Influenza viral challenge delivered directly to the respiratory tract within 1 year prior to challenge.
* History of adverse reaction to neuraminidase inhibitors e.g. oseltamivir
* Presence of any febrile illness or symptoms of upper viral respiratory infection:

  i. On the day of challenge/exposure or between admission for Influenza challenge/exposure and administration of the challenge inoculums (Donors) or exposure event (Recipients). Such subjects may be re-evaluated for enrollment in later studies after resolution of the illness; ii. Within 2 weeks prior to challenge or if challenge is set to occur during November, December, January, February, or March if there are any symptoms suggestive of viral respiratory infection occurring between screening and challenge.
* History of epistaxis (nose bleeds) more than 1 episode a month.
* Presence of household member or close contact (for an additional two weeks after discharge from the isolation facility) who is: (a) less than 3 years of age; (b) any person with any known immunodeficiency; (c) any person receiving immunosuppressant medications; (d) any person undergoing or soon to undergo cancer chemotherapy within 28 days of challenge; (e) any person who has diagnosed emphysema or COPD, is elderly residing in a nursing home, or with severe lung disease or medical condition including but not exclusive to the conditions listed in Appendix 4; or (f) any person who has received a transplant (bone marrow or solid organ).
* Any laboratory test which is abnormal and which is deemed by the Investigator to be clinically significant. (This includes blood chemistry, haematology, cardiac iso-enzymes, or urinalysis).
* Known IgA deficiency, immotile cilia syndrome, or Kartagener's syndrome.
* History of seasonal hay fever or a seasonal allergic rhinitis (SAR), including the use of symptomatic prescription only medication and non prescription medication.
* As a result of the medical interview, physical exam, or screening investigations, the Investigator considers the subject unfit for the study.
* Those employed or immediate relatives of those employed at Retroscreen Virology Ltd or the study site.
* Staff and students working directly in or for any of the Units in which the principal or a co-Investigator works.
* Immediate relatives of any of the principal or co-Investigators.
* Receipt of a northern hemisphere seasonal influenza vaccine in the 2006/07/08 winter seasons.
* Receipt of any systemic cytotoxic chemotherapy agent at any time.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
One or more individuals who develop a symptomatic illness confirmed as influenza A | 24 hourly

CONTACTS AND LOCATIONS:
Overall Officials: JONATHAN VAN-TAM, MD, Principal Investigator — University of Nottingham
Locations (1):
- Retroscreen Virology Ltd, London, United Kingdom

REFERENCES:
- See also: Related Info — http://www.flucamp.com